CLINICAL TRIAL: NCT02397369
Title: Comparative Evaluation of Efficacy of Different Methods of Tobacco Cessation Interventions Among BEST Employees in Mumbai : A Randomized Controlled Trial
Brief Title: Evaluation of Efficacy of Different Methods of Tobacco Cessation Interventions Among BEST Employees in Mumbai
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Gauravi Ashish Mishra, Associate Professor & Physician, Tata Memorial Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: TMHPOBEST2015
Record Dates: First submitted 2015-03-02; First posted 2015-03-24 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Compliance; Tobacco Use Cessation
Keywords: Education and evaluate post intervention KAP
MeSH Terms: conditions — Patient Compliance; Tobacco Use Cessation | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Tobacco users: Self Help (Experimental): Self-help intervention is defined as any manual or programme to be used by individuals to assist a quit attempt not aided by counsellors or group support.They include written materials on the health effects of tobacco, audio-or video tape or computer programmes.
  Interventions: Other: Tobacco users: Self Help
- Tobacco users:Telephonic counseling (Experimental): Telephone counseling is a way of providing individual counseling via telephone conversation or telephone hotlines. It can be proactive or reactive.
  Interventions: Behavioral: Tobacco users:Telephonic counseling
- Tobacco users:Behavioural therapy Only (Experimental): Behavioural therapy includes multiple sessions of Focus Group Discussion (FGD) and individual tobacco cessation counseling sessions. The participants in this group will be given advice to quit tobacco via multisession formal cognitive-behavioural therapy as per the Tobacco Cessation Clinic (TCC) guidelines.
  Interventions: Behavioral: Tobacco users:Behavioural therapy Only
- Tobacco users:Pharmacologic (Experimental): Pharmacotherapy in the form of Nicotine Replacement Therapy based on individual need assessment to relieve withdrawal symptoms in tobacco users when trying to quit.
  Interventions: Behavioral: Tobacco users:Behavioural therapy Only; Other: Tobacco users:Pharmacologic

INTERVENTIONS:
Other: Tobacco users: Self Help — This group will be given pictorial material and minimal written materials/ pamphlets describing health hazards of smokeless forms of tobacco and tips on tobacco cessation in general. The material will be interactively tailored to individual tobacco consumption characteristics and they will be followed up after 12 months.
  Other Names: Self help
  Arms: Tobacco users: Self Help
Behavioral: Tobacco users:Telephonic counseling — This group will be given proactive as well as reactive counseling. Medical social workers will proactively call all participants regularly and offer tobacco cessation counseling. In addition, they will call those participants who have planned their quit dates. Dedicated independent mobile numbers with 12 hours help lines will be made available to the participants to maximise the level of support. It will be scheduled in response to the needs to answer any type of help pertaining to quitting tobacco.
  Other Names: Telephonic
  Arms: Tobacco users:Telephonic counseling
Behavioral: Tobacco users:Behavioural therapy Only — 1. Focus Group discussion:
     This tobacco cessation intervention session will involve thirty minutes of focus group discussion with group behavioral therapy in groups of 5-10 individuals for reinforcement of tobacco use prevention and cessation advice. Group discussion is intended to improve understanding by exploring, sharing and reflecting psychosocial, familial, environmental issues which attribute to the problem.
  2. Individual tobacco cessation counseling sessions:
  Individual counseling is commonly used to help people who are trying to quit tobacco. The counseling adopting an interactive problem-solving approach will be done by trained Medical Social Workers providing face-to-face sessions for 10-15 minutes per participant.
  Arms: Tobacco users:Behavioural therapy Only; Tobacco users:Pharmacologic
Other: Tobacco users:Pharmacologic — Pharmaco Therapy will consist of:
  Nicotine Chewing Gums:
  Dose: 2 mg/4 mg, 10-15 pieces per day with maximum dose of 24 pieces/day depending on cravings Total Duration: 12 weeks Duration of treatment: Higher dose for 4-6 weeks, with weaning till 2-3 months Side effects: Bad taste, Throat irritation, burning in mouth, nausea, vomiting, hiccups, increased heart beat etc
  Nicotine Transdermal patches:
  Dose: 7 mg/10 mg/14 mg/21 mg -for 24-hours use. Total Duration: 12 weeks Duration of treatment: Higher strength patch for 2 weeks and depending on cravings will be gradually decreased till 4 weeks Side effects: Skin irritation, dizziness, sleep problems, increased heart beat etc
  Other Names: Drug
  Arms: Tobacco users:Pharmacologic

SUMMARY:
Tobacco use is the single most preventable cause of premature adult death globally. It is one of the major causes of death and disease in India, accounting for nearly 0.9 million deaths every year.

Bombay Electric Supply and Transport (BEST), one of the biggest public transport undertaking in Mumbai City, has imposed a ban on tobacco use in public transport buses and under Motor Vehicle Act has empowered the drivers and bus conductors to take suitable action against commuters found to be using tobacco. However in addition to commuters using tobacco in the BEST premises, large number of bus drivers and conductors are known to use tobacco on the job. There are various approaches to a tobacco cessation programme, like behavioural therapy, pharmacotherapy, providing self help material, telephone counseling, quit lines etc.

Hence in terms of the workplace environment, understanding the factors leading to tobacco use maintenance and the effective approaches for cessation is of critical importance for formulating workplace tobacco prevention and cessation interventions that are applicable to transport work employee settings. The success of these methods needs to be comparatively evaluated among the different forms of tobacco users. Hence, the present study will be undertaken with the following objectives:

DETAILED DESCRIPTION:
RESEARCH OBJECTIVES:

1. To study the Knowledge, Attitudes and Practices (KAP) regarding tobacco among BEST employees in Mumbai
2. To study the occupational correlates of tobacco consumption across various grades of BEST employees
3. To educate them regarding hazards of tobacco.
4. To offer BEST employees Preventive Oncology screening facilities and evaluate the compliance for screening and determine the rate of oral pre-cancers.
5. To study the post-intervention KAP regarding tobacco
6. To randomly assign the BEST employees using tobacco to one of the four tobacco cessation interventions and study the compliance to the same.
7. To determine the rate of tobacco cessation after twelve months of follow-up.
8. To comparatively evaluate the success of the four approaches of tobacco cessation, viz. providing self help material, telephone counseling, behavioural therapy and behavioural + pharmacotherapy, among users of different forms of tobacco.

Methodology:

Study Design: Four arm interventional study

Step 1: Around 4000 BEST employees in Mumbai will be enrolled after explaining the programme and obtaining informed consent. They will be interviewed with the help of a well structured questionnaire to collect information about their Knowledge, Attitudes and Practices (KAP) regarding tobacco, their attitudes and experiences regarding smoke free public places with specific reference to smoke free BEST buses.

Step 2: The BEST employees will be given detailed health education regarding hazards of tobacco and the need for smoke free BEST buses. The BEST employees will be invited to participate in Preventive Oncology (PO) screening (mainly oral cancer screening).

Step 3: The BEST employees will be again interviewed with the help of a well structured questionnaire to collect information of their post-intervention KAP regarding tobacco and smoke free public places.

Step 4: The BEST employees using tobacco will be registered at the Tobacco cessation clinic and will be invited to participate in the first session of tobacco cessation counseling.

The BEST employees using smoking forms of tobacco will be offered interventions and will be followed up as per the TCC protocol.

The smokeless tobacco users will be randomly assigned into one of the four groups to receive intervention. Each group of employee will receive one of the four interventions as follows: self help material, telephone counseling, behavioural therapy and behavioural + pharmacotherapy.

The pharmacotherapy intervention in the form of Nicotine Replacement Therapy comprising of Nicotine chewing gums or patches (Transdermal patches) will be based on individual need assessment to relieve withdrawal symptoms in tobacco users when trying to quit.

Nicotine Chewing Gums:

Dose: 2 mg/4 mg, 10-15 pieces per day with maximum dose of 24 pieces/day depending on cravings Total Duration: 12 weeks Duration of treatment: Higher dose for 4-6 weeks, with weaning till 2-3 months Side effects: Bad taste, Throat irritation, burning in mouth, nausea, vomiting, hiccups, increased heart beat etc

Nicotine Transdermal patches:

Dose: 7 mg/10 mg/14 mg/21 mg -for 24-hours use. Total Duration: 12 weeks Duration of treatment: Higher strength patch for 2 weeks and depending on cravings will be gradually decreased till 4 weeks Side effects: Skin irritation, dizziness, sleep problems, increased heart beat etc

Step 5: The BEST employees with lesions will be followed up at the Preventive Oncology screening clinic as per PO protocols. The tobacco users enrolled in the TCC will be followed up over a period of twelve months with three interventions in between and a post-intervention follow-up.

Variables to be estimated:

1. Knowledge, Attitudes and Practices (KAP) regarding tobacco among BEST employees.
2. The compliance for availing the services at Preventive Oncology screening facilities and Tobacco cessation clinic at the Tata Memorial Hospital
3. The rate of oral pre-cancers among BEST employees.
4. The post-intervention KAP regarding tobacco.
5. The rate of tobacco cessation after one year follow-up.
6. Compare the success of various approaches for tobacco cessation and assess the compliance for the same.

Data Analysis:

Data entry will be done in the Department of Preventive Oncology, Tata Memorial Hospital using Statistical Package for Social Sciences (SPSS) version 18. Checks for consistency, data safety and analysis will be carried out at regular intervals. Both descriptive and inferential statistics will be generated for describing variables under the study objectives.

ELIGIBILITY:
Inclusion Criteria:

* BEST employees in Mumbai

Exclusion Criteria:

* BEST employees not willing to give consent

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2015-03; Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Knowledge, Attitudes and Practices (KAP) regarding tobacco among BEST employees. | 60 months
  To study the Knowledge, Attitudes and Practices (KAP) regarding tobacco among BEST employees in Mumbai

OTHER OUTCOMES:
Compliance for availing the services at Preventive Oncology screening facilities and Tobacco cessation clinic at the Tata Memorial Hospital | 60 months
  randomly assign the BEST employees using tobacco to one of the four tobacco cessation interventions and study the compliance to the same.
Rate of oral pre-cancers among BEST employees | 60 months
  To assesses rate of precancer among BEST employees
Rate of tobacco cessation after one year follow-up | 60 months
  . To determine the rate of tobacco cessation after twelve months of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Gauravi A Mishra, Assoc Prof, Principal Investigator — Tata Memorial Hospital, Mumbai; Sharmila A Pimple, Professor, Principal Investigator — Tata Memorial Hospital, Mumbai
Locations (1):
- Tata Memorial Hospital, Parel, Mumbai, Maharashtra, India